CLINICAL TRIAL: NCT06689150
Title: Evaluation of the Contraceptive Efficacy, and Safety of Different Types of Progestron Only Pills (Drosperinon 4 mg, Desogestrel 75 pg and Levonorgestrel 30 pg), A Comparative Randomized Controlled Trial
Brief Title: Evaluation of the Contraceptive Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Heba Tullah Mohamed Alsyed, Resident of Obstetrics & Gynecology, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hebatu Allah Mohamed
Record Dates: First submitted 2024-10-25; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2023-08

CONDITIONS: Menstrual Bleeding, Heavy
Keywords: Drospirenon; Desogestrel; Levonorgestrel
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Drospirenon (drospinetta) (Active Comparator): About 100 women took Drospirenon (drospinetta) tab every day 24 and 4 placipo tablets for four days
  Interventions: Drug: Drospinetta
- Group B: Desogestrel (Cirazette) (Active Comparator): About 100 women took Desogestrel (Cirazette) tablet every day
  Interventions: Drug: Drospinetta
- Group C: Levonorgestrel (Microlute) (Active Comparator): About 100 women took Levonorgestrel (Microlute) tablet every day
  Interventions: Drug: Drospinetta

INTERVENTIONS:
Drug: Drospinetta — To evaluate the three different types of POPs, the new POPs Drosperinon 4 mg, Desogestrel 75 pg, and Levonorgestrel 30 pg in healthy female subjects as regard to the contraceptive efficacy, bleeding pattern, acceptability and safety
  Other Names: Cirazette; Micrlute

SUMMARY:
Combined oral contraceptives are not the preparation of first choice in breastfeeding women as they may influence the quality and quantity of breast milk. In these cases, a progestogen-only pill is a suitable alternative, since progestogen-only pills contain no estrogen at all and a much lower dose of progestogen than do combined oral contraceptives

Therefore, progestogen-only pills may also be more acceptable than combined oral contraceptives to women suffering from medical conditions that are associated with the use of combined oral contraceptives (e.g. nausea, headache and breast tension).

DETAILED DESCRIPTION:
The most widely prescribed form of hormonal contraception is the combined oral contraceptive, which offers good contraceptive efficacy and a number of non-contraceptive benefits.

However, the combined pill has also been associated with some adverse effects, mainly related to the vascular system, i.e. a slightly higher risk of venous thromboembolic events .

Most studies have linked the risk of venous thromboembolic events dose dependently to the estrogen component. Estrogen-containing oral contraceptives may, therefore, be contraindicated in women with risk factors for venous thromboembolic events.

The current progestogen-only pills contain levonorgestrel, norethisterone, lynestrenol or ethynodiol diacetate have a multifaceted, mode of action .

Ovulation inhibition is achieved in about half of the cycles and contributes only partly to the effectiveness of the method, with effects on the cervical mucus and the endometrium, thus providing additional contraceptive reliability .

Drawbacks of the traditional progestogen-only pills in comparison to COCs are the high incidence of irregular bleeding, the higher rate of ectopic pregnancies and a slightly lower contraceptive efficacy. If a newly developed progestogen-only pill improves on one or more of these drawbacks, it may be a valuable addition to the traditional progestogen-only pills .

Levonorgestrel, also known as the morning-after pill, is a first-line oral emergency contraceptive pill with approval from the World Health Organization to prevent pregnancy. It is FDA-approved to be used within 72 hours of unprotected sexual intercourse or when a presumed contraceptive failure has occurred .

Desogestrel is a selective progestogen with a lower androgenic activity than the progestogens used in the traditional progestogen-only pills. Therefore, a dose that is high enough to obtain inhibition of ovulation is not likely to trigger androgen-related side-effects. Levonorgestrel is a second-generation synthetic progestogen that is the active component of the racemic mixture of norgestrel. It binds to progesterone and androgen receptors, where it can delay gonadotropin-releasing hormone from being released from the hypothalamus .

Drospirenone is a synthetic spironolactone analogue and progestin with progestational and anti-mineralocorticoid activity. Drospirenone binds to the progesterone receptor; the resulting complex becomes activated and binds to specific sites on DNA. This results in a suppression of LH activity and an inhibition of ovulation as well as an alteration in the cervical mucus and endometrium. This leads to an increased difficulty of sperm entry into the uterus and implantation. This drug is used in oral contraceptives.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 45 years.
* Non obese women with BMI between 18.5 : 29.9 kg/m2.
* Healthy women with good physical and mental health.
* Sexually active.
* Women have normal cycles (regular interval, duration, and amount of bleeding.
* Women willing to accurately fill in the diary card with daily information on vaginal bleeding and pill intake
* Women willing to give written informed consent.

Exclusion Criteria:

* obese medical history
* Contraindications to the use of progesterone only pills with medical eligibility criteria mec category 3 or 4: (malabsorptive procedures, current or history of ischemic heart disease, history of cerebrovascular accident, systemic lupus erythematosus, breast cancer, cirrhosis, liver tumors or antimicrobial therapy).
* Women with allergy from study medications.
* Women refusing to participate in the study.

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Irregular Vaginal Bleeding | 9 Months
  Efficacy of the different types of the progesterone only pills as : (Drosperinon tablets, Desogestrel tablets and Levonorgestrel tablets) which will be initiated on the first day of menstruation in controlling of irregular vaginal bleeding during menses

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ali Mohamed Nasr, M.D, Study Chair — Al-Azhar University, Assuit
Locations (1):
- Al-Azhar University Hospitals, Asyut, Egypt